CLINICAL TRIAL: NCT03731312
Title: Variability of Daily Iodine Intake: The Effects of Intra- and Inter-individual Variability on Estimated Intake in Iodine Nutrition Studies
Brief Title: Variability of Daily Iodine Intake: The Effects of Intra- and Inter-individual Variability in Iodine Nutrition Studies
Acronym: VIOLET
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: VIOLET
Record Dates: First submitted 2018-10-01; First posted 2018-11-06 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Iodine Deficiency
Keywords: Iodine; Urinary iodine concentration

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, Dried blood spot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: We will collect two repeated spot urine samples, a DBS sample and obtain weight in all 600 study participants. In a randomly selected subsample (n=200) a third repeat spot urine sample and one 24 h urine will additionally be collected.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study and no interventions will be administered.

SUMMARY:
Iodine status in populations is assessed using urinary iodine concentration (UIC) measured in spot urine samples. The iodine intake is classified as deficient, sufficient, or excessive iodine based on the median UIC (mUIC). However, this approach has limitations, as it does not quantify the prevalence of individuals with habitually deficient or excess iodine intakes. The EAR cut-point method has the potential to quantify prevalence of iodine deficiency and excess. However, little is known about the effects of the inter- and intra-individual variance of UIC.

The aim of the study is to quantify the intra-individual variability in dietary iodine intake. The overall goal is to estimate the prevalence of iodine deficiency and excess in the study population and propose sample size recommendations for future iodine nutrition population studies. The results will provide evidence guiding international recommendations for iodine nutrition studies.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* Non-lactating
* Non-smoking
* Residence in Switzerland ≥12 months
* Generally healthy
* No family history of goiter
* No exposure to iodine containing contrast agents during the last 12 months - Informed consent given

Exclusion Criteria:

* Participant is not able to understand the study information or procedure, e.g. due to linguistic barriers

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women of reproductive age and residents of Switzerland since at least 12 months
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Estimated daily urinary iodine excretion | 7 days
  Estimated urinary iodine excretion (µg/day) will be obtained from urinary iodine concentration (UIC) and urinary creatinine concentration (UCC) measured in two repeat spot urine samples collected within 7 days

SECONDARY OUTCOMES:
Measured daily iodine excretion | 1 day
  Measured daily iodine excretion (µg/day) will be obtained from urinary iodine concentration (UIC) and urine volume in a 24 h urine collection
Thyroid function test TSH | 1 day
  TSH concentration (mU/L) measured in dried blood spots
Thyroid function test total T4 | 1 day
  Total T4 concentration (nmol/L) measured in dried blood spots
Thyroid function test Tg | 1 day
  Tg concentration (µg/L) measured in dried blood spots

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Rigutto-Farebrother, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arns-Glaser L, Zihlmann R, Gessler S, Verkaik-Kloosterman J, Zandberg L, Assey VD, Rigutto-Farebrother J, Braegger CP, Zimmermann MB, Andersson M. Estimating habitual iodine intake and prevalence of inadequacy from spot urine in cross-sectional studies: a modeling analysis to determine the required sample size. Am J Clin Nutr. 2023 Jun;117(6):1270-1277. doi: 10.1016/j.ajcnut.2023.03.012. Epub 2023 May 4. PMID 37270291